CLINICAL TRIAL: NCT04070547
Title: The Effect of Transcutaneous Vagus Nerve Stimulation on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: COG-STIM
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Function
Keywords: Cognitive function; transcutaneous vagal nerve stimulation; autonomic nervous system; cognitive health/impairment

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of 4 groups - receiving either transcutaneous vagal nerve stimulation or sham in first 2 weeks (Early group), or being first 2 weeks on the waiting list and receiving either transcutaneous vagal nerve stimulation or sham in the second 2 weeks of the study participation (Late group). The randomization will have two steps: 1.) Prior to the first laboratory session all participants will be assigned into either Early or Late group; 2.) At the end of the pre-intervention laboratory session participants will be randomized between tVNS or sham stimulation.
Who Masked: Participant
Masking Description: The sham stimulation experience is very similar to the tVNS stimulation experience. Participants will be provided a detailed instructions and manual how to use the tVNS device and at what part of the ear they will place the electrode on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early tVNS (Experimental): First 2 weeks this group will receive transcutaneous vagal nerve stimulation 4 hours a day (day 1 to day 14). Then participants will be followed for another 2 weeks (day 15 to day 28) without any intervention. Laboratory testing will be carried out three times with average of 14 days between sessions: on day 1 (pre-intervention), on day 14 (post-intervention) and on day 28 (follow-up).
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Early Sham (Experimental): First 2 weeks this group will receive sham stimulation 4hours a day (day 1 to day 14). Then participants will be followed for another 2 weeks (day 15 to day 28). Laboratory testing will be carried out three times with average of 14 days between sessions: on day 1 (pre-intervention), on day 14 (post-intervention) and on day 28 (follow-up).
  Interventions: Device: Sham stimulation
- Late tVNS (Experimental): First 2 weeks this group will be on a waiting list (day 1 to day 14). Then participants will receive transcutaneous vagal nerve stimulation 4hours a day (day 15 to day 28). Laboratory testing will be carried out three times with average of 14 days between sessions: on day 1 (waiting), on day 14 (pre-intervention) and on day 28 (post-intervention).
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Late Sham (Experimental): First 2 weeks this group will be on a waiting list (day 1 to day 14). Then participants will receive sham stimulation 4hours a day (day 15 to day 28). Laboratory testing will be carried out three times with average of 14 days between sessions: on day 1 (waiting), on day 14 (pre-intervention) and on day 28 (post-intervention).
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — Non-invasive stimulation provided by transcutaneous electrical nerve stimulation device 4hours a day at 25Hz, 250 μs pulse width placed on tragus.
  Arms: Early tVNS; Late tVNS
Device: Sham stimulation — Sham stimulation will be performed using electrodes 4 hours a day placed on earlobe.
  Arms: Early Sham; Late Sham

SUMMARY:
Cognitive health is generally considered a key component of quality of life. Current evidence indicates that a large number of individuals are at a high risk for cognitive impairment from many causes as they age. In order to preserve and enhance positive out-comes by targeted efficient preventive and therapeutic strategies it is important to understand potential mechanisms and predictors of cognitive health and impairment. Withdrawal of vagal (parasympathetic) activity has been proposed as one of the biological pathways involved in cognitive impairment. Transcutaneous vagus nerve stimulation (tVNS) has shown potential as a noninvasive and safe therapeutic treatment due to its direct influence on brain systems involved in cognition. However, the role of vagal modulation in cognitive functioning and impairment and the influence of tVNS, particularly long-term tVNS, on cognition are not yet completely understood. Here the investigators aim to investigate the effect of long-term (14days) intensive transcutaneous vagus nerve stimulation on cognitive functions in relatively healthy young-to-older adults.

DETAILED DESCRIPTION:
Cognitive health is generally considered a key component of quality of life. Current evidence indicates that a large number of individuals are at high risk for cognitive impairment from many causes as they age. In order to preserve and enhance positive cognitive health outcomes by targeted efficient preventive and therapeutic strategies, it is important to understand potential mechanisms and predictors of cognitive health and impairment. Withdrawal of vagal (parasympathetic) activity has been proposed as one of the biological pathways involved in cognitive impairment. Transcutaneous vagus nerve stimulation (tVNS) has shown potential as noninvasive and safe therapeutic treatment due to its direct influence on brain systems involved in cognition. However, the role of vagal modulation in cognitive functioning and impairment and the influence of tVNS, particularly long-term tVNS, on cognition are not yet completely understood. Here the investigators aim to investigate the effect of long-term (14days) intensive transcutaneous vagus nerve stimulation on cognitive functions in relatively healthy young-to-older adults.

Little work has been done investigating the effect of long-term tVNS in healthy men and women. In light of preventive medicine, the question is whether increased vagus nerve modulation and long-term tVNS improve memory and executive functioning and potentially help to prevent healthy person vulnerable to cognitive impairment from manifesting cognitive deficits. Or if they can slow down the process of cognitive aging inevitable for every human being.

ELIGIBILITY:
Inclusion Criteria:

* relatively healthy adults

Exclusion Criteria:

* cardiovascular disease (e.g. arythmia, history of coronary heart disease, history of stroke),
* severe mental condition (e.g. significant depression, schizophrenia, autism, significant anxiety disorder)
* severe neurological condition (e.g. epilepsy, brain tumors, significant migraine, traumatic brain injury)
* brain surgery
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Rey´s Auditory Verbal Learning Test | 12 minutes
  Test of short-term memory, learning and recall to assess delayed memory
Flanker test | 4 minutes
  Test that measures attention and executive function specifically response inhibition
Set Shifting | 7 minutes
  Test of executive function specifically cognitive flexibility
N-back and 2N-back | 10 minutes
  Test of executive function specifically working memory
Random number generation | 5 minutes
  Test of executive function specifically cognitive flexibility
Emotion Recognition Task | 5 minutes
  Test of emotion recognition
Emotion GoNoGo | 5 minutes
  Test of emotion inhibition and emotion regulation

SECONDARY OUTCOMES:
Supine and task dependent heart rate variability | 63 minutes
  These tests will measure supine resting heart rate variability and changes in heart rate variability during each cognitive challenge task (memory, executive function and emotion regulation tests).

CONTACTS AND LOCATIONS:
Overall Officials: Vera Jandackova, Principal Investigator — University of Ostrava
Locations (1):
- University of Ostrava, Faculty of Medicine, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: Undecided